CLINICAL TRIAL: NCT01000571
Title: Immunogenicity and Safety of Inactivated H1N1 Swine-origin Influenza Monovalent Vaccine in Immunocompromised Children and Young Adults
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SOVAC
Record Dates: First submitted 2009-10-19; First posted 2009-10-23 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: H1N1 Pandemic Flu
Keywords: H1N1 pandemic flu

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection will be done according to the description provided in the institutional policy manual. When possible, blood draws will be made through existing implanted catheters. If the research participant does not have a catheter, a peripheral venipuncture will be performed. Serum and whole blood for immune assays will be frozen at -20ºC or in liquid nitrogen until processed in batched assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- H1N1 pandemic influenza vaccine recipient: Children and young adults between the ages of 6 months and 21 years and 13 kg or greater in body weight with underlying conditions of cancer, HIV, sickle cell disease or receipt of a stem cell transplant more than a year prior to study entry and who will receive inactivated H1N1 swine-origin monovalent influenza vaccine in the winter/fall of 2009-2010 as part of their routine clinical care.Target total accrual of up to 400 children and young adults stratified based on their underlying diagnosis as follows: 150 children or young adults with cancer, 100 with human immunodeficiency virus (HIV), 100 with sickle cell disease, and 50 with receipt of a stem cell transplant more than a year prior to study entry.

SUMMARY:
This study will evaluate the immunogenicity and safety of inactivated H1N1 swine-origin monovalent influenza vaccine in immunocompromised children and young adults.

DETAILED DESCRIPTION:
This is a prospective observational study. This study will not dictate vaccine administration, nor the vaccine product to be used. It will collect data in St Jude patients who will receive the vaccine as part of their clinical care per institutional guidelines. Research participants will receive two doses of inactivated H1N1 swine-origin monovalent influenza vaccine administered 28 days apart as part of clinical care. Each dose contains 15 mcg of hemagglutinin antigen (HA).Follow-up visits will be scheduled 28 days after each dose and at day 208+/- 14 days for blood work. The day of administration of the first vaccine dose is counted as day 0. At each of these visits, blood will be collected to assess for immunogenicity. Research participants will be given a diary card to record symptoms for 28 days . They will be asked to bring this diary back at the next visit. Other vaccine-related adverse events will also be collected by retrospective chart review.

Children and young adults between the ages of 6 months and 21 years and 13 kg or greater in body weight who have an underlying diagnosis of cancer, HIV, sickle cell disease or receipt of a stem cell transplant more than a year prior to study entry and who will receive inactivated H1N1 swine-origin monovalent influenza vaccine in the winter/fall of 2009-2010 as part of their routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months through 21 years of age at the time of entry into the study;
* Body weight of 13 kg or greater at the time of entry into the study;
* Participant is immunocompromised due to cancer, HIV, or sickle cell disease or receipt of a stem cell transplant;
* Participant or participant's parent/legal guardian available by telephone during the course of the study;
* Written informed consent (and assent, if applicable) obtained;
* Potential research participant received or will receive H1N1 swine-origin monovalent influenza vaccine within 24 hours of study entry.

Exclusion Criteria:

* Proven history, by RT-PCR, of H1N1 swine-origin influenza infection prior to study entry;
* Receipt of a stem cell transplant within one year prior to study entry;
* Participation in P1088 study.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults between the ages of 6 months and 21 years and 13 kg or greater in body weight who have an underlying diagnosis of cancer, HIV, sickle cell disease or receipt of a stem cell transplant more than a year prior to study entry and who will receive inactivated H1N1 swine-origin monovalent influenza vaccine in the winter/fall of 2009-2010 as part of their routine clinical care. Stem cell transplant recipients in the first year following their transplant are excluded.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
This study will document Seroprotection (a post-vaccine antibody response ≥ an HI titer of 1:40). | 1.5 years

SECONDARY OUTCOMES:
This study will document seroconversion rates (a 4-fold or greater rise in HI titer comparing pre- and post-vaccine sera). | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hana Hakim, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St.Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org